CLINICAL TRIAL: NCT03271424
Title: Innovations in HIV Testing to Enhance Care for Young Women and Their Peers and Partners
Brief Title: Innovations in HIV Testing (TI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Witwatersrand, South Africa (Other); University of California, San Francisco (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 15-1361a; 5R01HD083033 (NIH)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Qualitative focus group discussions (FGDs) with male and female community members aged 18 - 24
  In-clinic observation of HIV self-testing and completion of a brief CAPI/ACASI interview with male and female community members aged 18 - 24
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Focus Group Discussions (No Intervention): Focus group discussions (FGD) with young women (n=2 FGDs) and young men (n=2 FGDs) in the study area to determine the best way to offer self-testing to study participants.
- In Clinic Observation-Both (Active Comparator): 10 young women and 10 young men were assigned and conducted BOTH of the HIV self-tests. Participants tried two different self-testing kits, one that is oral fluid based (saliva), Oraquick HIV Self Test, and one that is blood based via a finger prick, Atomo HIV Self Test. Oraquick HIV Self Test and Atomo HIV Self Test - Both
  Interventions: Diagnostic Test: Oraquick HIV Self Test and Atomo HIV Self Test - Both
- In Clinic Observation-Subject Choice (Active Comparator): 20 young women and 20 young men were assigned and conducted EITHER of the HIV self-tests. Investigators asked them to choose which test they would prefer to use, one that is oral fluid based (saliva), Oraquick HIV Self Test, or one that requires the use blood via a finger prick, Atomo HIV Self Test. Oraquick HIV Self Test - Choice; Atomo HIV Self Test - choice
  Interventions: Diagnostic Test: Oraquick HIV Self Test - Choice; Diagnostic Test: Atomo HIV Self Test - Choice

INTERVENTIONS:
Diagnostic Test: Oraquick HIV Self Test - Choice — This is an oral swab in home HIV test.
  Arms: In Clinic Observation-Subject Choice
Diagnostic Test: Atomo HIV Self Test - Choice — This is a blood finger prick in home HIV test.
  Arms: In Clinic Observation-Subject Choice
Diagnostic Test: Oraquick HIV Self Test and Atomo HIV Self Test - Both — This is an oral swab in home HIV test and this is a blood finger prick in home HIV test.
  Arms: In Clinic Observation-Both

SUMMARY:
The investigators propose to improve HIV prevention and care through expanding HIV testing options to include self-testing for young women, their peers and their sex partners, and by facilitating linkage to care.

DETAILED DESCRIPTION:
Study Description Brief Summary: The investigators propose to improve HIV prevention and care through expanding HIV testing options to include self-testing for young women, their peers and their sex partners, and by facilitating linkage to care.

Detailed Description: The investigators propose to improve HIV prevention and care through expanding HIV testing options to include self-testing for young women, their peers and their sex partners, and by facilitating linkage to care. In this study the investigators proposed two phases. The first phase, explained in this submission, is formative and involved two parts: 1) conducting formative qualitative research to understand perceptions of HIV testing and HIV self-testing in the study population and 2) conducting observed HIV self-testing to better understand any challenges with self-testing and the materials needed to make the process clear. The second phase of the study is a randomized controlled trial where the investigators will randomize approximately 400 young women to receive either 1) CHOICE of self-testing or clinic-based HIV Counseling and Testing (HCT) or 2) clinic based HCT. Once young women have been randomized, they will be asked to recruit up to 4 peers or male sex partners to test with the method of their randomization group.

ELIGIBILITY:
FGD Inclusion Criteria:

* Females and males aged 18 - 24
* Able and willing to provide informed consent
* Residing in the selected villages

Observation Inclusion Criteria:

* Females and males aged 18 -24
* Able and willing to provide informed consent
* Residing in the selected villages
* Not known to be HIV positive (not reporting a previous positive test)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Enrolled participants need to self-identify as female or female for their respective data collection.
Enrollment: 95 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Pettifor, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Medical Research Council/Wits University Rural Public Health and Health Transitions Research Unit, Agincourt, Mpumalanga, South Africa

RESULTS

PARTICIPANT FLOW:
Period: November 2015
Arm/Group | In Clinic Observation-Both | Focus Group Discussions | In Clinic Observation-Subject Choice
Started | 20 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 0 | 0 | 0
Period: December 2015
Arm/Group | In Clinic Observation-Both | Focus Group Discussions | In Clinic Observation-Subject Choice
Started | 0 | 35 | 0
Completed | 0 | 35 | 0
Not Completed | 0 | 0 | 0
Period: April-May 2016
Arm/Group | In Clinic Observation-Both | Focus Group Discussions | In Clinic Observation-Subject Choice
Started | 0 | 0 | 40
Completed | 0 | 0 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Focus Group Discussions | In Clinic Observation-Both | In Clinic Observation-Subject Choice | Total
Number analyzed (Participants) | 35 | 20 | 40 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 20 | 40 | 95
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 20 [18 to 24] | 20 [18 to 24] | 20 [18 to 24] | 20 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 20 | 46
  Male | 19 | 10 | 20 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 35 | 20 | 40 | 95

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Summaries of Participant Experience in Focus Group Discussions
Description: Qualitative Summaries for recruitment of peers/sex partners, issues related to privacy and spaces for testing, options for post-test counseling, optimizing return visits, and preferences for contact
Time Frame: 6 months post study start
Measure: Number; unit: number of times reported in FGD
Arm/Group | Focus Group Discussions
Number analyzed (Participants) | 35
number of times reported in FGD
  HIV Self Test (HST) Acceptability | 100
  HST Context | 7
  HST Kit Preference | 26
  HST motivation | 10
  HST Recommendations | 29
  Supportive resources | 12

2. Primary Outcome: Quantitative Summaries of Participants Experience in Observation Sessions
Description: Frequency counts of clarity of instructions, comfort using the test, confidence in test result, difficulty performing the test and reading results
Time Frame: 12 month post study start
Measure: Count of Participants; unit: Participants
Groups:
- In Clinic Observation-Both (Oraquick Results); In Clinic Observation - Both (Atomo Results): 10 young women and 10 young men were assigned and conducted BOTH of the HIV self-tests. Participants tried two different self-testing kits, one that is oral fluid based (saliva), Oraquick HIV Self Test, and one that is blood based via a finger prick, Atomo HIV Self Test. Oraquick HIV Self Test and Atomo HIV Self Test - Both
  Oraquick HIV Self Test and Atomo HIV Self Test - Both: This is an oral swab in home HIV test and this is a blood finger prick in home HIV test.
- In Clinic Observation-Subject Choice (Oraquick Results); In Clinic Observation-Subject Choice (Atomo Results): 20 young women and 20 young men conducted EITHER of the HIV self-tests. Investigators asked them to choose which test they would prefer to use, one that is oral fluid based (saliva), Oraquick HIV Self Test, or one that requires the use blood via a finger prick, Atomo HIV Self Test. Oraquick HIV Self Test - Choice; Atomo HIV Self Test - choice
  Oraquick HIV Self Test - Choice: This is an oral swab in home HIV test.
  Atomo HIV Self Test - Choice: This is a blood finger prick in home HIV test.
Arm/Group | In Clinic Observation-Both (Oraquick Results) | In Clinic Observation - Both (Atomo Results) | In Clinic Observation-Subject Choice (Oraquick Results) | In Clinic Observation-Subject Choice (Atomo Results)
Number analyzed (Participants) | 20 | 20 | 32 | 8
Participants
  Found Instructions Clear | 19 | 19 | 30 | 8
  Were Very Comfortable Using the Test | 16 | 14 | 24 | 6
  Very Easy to use the Test | 18 | 13 | 27 | 7
  Very Easy to Interpret Results | 18 | 18 | 31 | 8

ADVERSE EVENTS:
Arm/Group | Focus Group Discussions | In Clinic Observation-Both | In Clinic Observation-Subject Choice
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/20 | 0/40
Other Adverse Events (participants affected / at risk) | 0/35 | 0/20 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes